CLINICAL TRIAL: NCT05771116
Title: Erector Spinae Catheter Versus Paravertebral Catheter for Pain Management in Modified Radical Mastectomy for Cancer Patients: A Randomized Double-Blind Non-inferiority Trial
Brief Title: Erector Spinae Catheter Versus Paravertebral Catheter for Postoperative Analgesia in Cancer Patients Post Mastectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2212-501-034
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An independent observer who will be blind to the group assignment checked the intraoperative and postoperative data also patient will be be blinded also
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erecto Spinae Plane Block group (Active Comparator): a high-frequency linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T7 spinous process. This should reveal three muscles superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. The skin will be anaesthetized using 3ml of 2% Lidocaine. A 20-gauge block needle will be inserted in-plane in a cephalad-to-caudad direction to place the tip into the fascial plane on the deep (anterior) aspect of erector spinaemuscle;20ml bupivacaine 0.25% will be injected. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process The needle will be removed and the catheter secured with adhesive.
  Interventions: Procedure: ERECTOR SPINAE PLANE BLOCK and PARAVERTEBRAL BLOCK:; Procedure: PARAVERTEBRAL BLOCK:
- the paravertebral group (Active Comparator): After identification of the transverse process, internal intercostal membrane (IIM), and pleura at the T3 and T6 levels, an out-of-plane needle guidance technique was used to perform the PVB.The success of both blocks will be confirmed by loss of pinprick sensation on the dermatomal site of the block
  •blocks will be activated ,After negative aspiration, 0.5 ml/kg 0.25% bupivacaine (max 20 ml) will be injected. Afterwards, a 20 gauge peripheral nerve catheter will be easily threaded into the space. The needle will be removed and the catheter secured with adhesive.
  Interventions: Procedure: ERECTOR SPINAE PLANE BLOCK and PARAVERTEBRAL BLOCK:; Procedure: PARAVERTEBRAL BLOCK:

INTERVENTIONS:
Procedure: ERECTOR SPINAE PLANE BLOCK and PARAVERTEBRAL BLOCK: — catheter will be placed for ERECTOR SPINAE PLANE BLOCK
Procedure: PARAVERTEBRAL BLOCK: — catheter will be placed for PARAVERTEBRAL BLOCK

SUMMARY:
All patients admitted in National Cancer institute, Cairo University for breast surgeries will be investigated for inclusion criteria in the current study. And will be enrolled if fulfilled the criteria into 2 groups

.70 patients will be included in this prospective randomized study. The patients will be allocated into two groups: the ESPB group (group E, n = 35) , and the paravertebral group (group P, n =35)

* All patients will do Ultrasound-guided ESPB for group E and PVB for group P before receiving general anesthesia
* Postoperatively Patients in both groups will receive intravenous morphine 3 mg as rescue analgesic

DETAILED DESCRIPTION:
* 70patients will be included in this prospective randomized study. The patients will be allocated into two groups: the ESPB group (group E, n = 35) , and the paravertebral group (group P, n =35)
* All patients will do Ultrasound-guided ESPB for group E and PVB for group P before receiving GA
* Postoperatively Patients in both groups will receive intravenous morphine 3 mg as rescue analgesic.
* Random numbers were generated using a computer-generated randomization code and were sealed in an opaque envelope. Randomization was conducted by a person who was not involved in the study.
* An independent observer who was blind to the group assignment checked the intraoperative and postoperative data.
* VAS pain score immediately postoperative and at 2,4,6, 8,12,18,24,36 ,48hrs.postoperative.

ELIGIBILITY:
Inclusion Criteria:

.Physical status ASA II.

. Patients (age 20-70yrs) scheduled for breast surgeries for breast cancer under general anesthesia

Exclusion Criteria:

.History of psychological disorders.

* Known sensitivity or contraindication to local anesthetics.
* Localized infection at the site of block.
* patients with coagulopathy or an (INR ≥ 2)

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female post mastectomy
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Total 48 hours Post-operative opioid consumption to keep VAS score ≤4. | 48 hours postoperative
  the VAS score rating, in which 0 = "no pain" and 10 = "worst possible pain". both during rest and movement

SECONDARY OUTCOMES:
1st request of analgesia | 48 hours postoperative
  1st request of analgesia , any hemodynamic instability and complications

CONTACTS AND LOCATIONS:
Overall Officials: suzan adlan, lecturer, Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- NCIEgypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No